CLINICAL TRIAL: NCT04301193
Title: Efficacy of Sonorheometry Point of the Care Device in Determining Low Fibrinogen Levels in Pregnant Blood: an Invitro Dilution and Reconstitution Study
Brief Title: Evaluation of Novel Point of Care Coagulation System in Pregnant Women
Acronym: CCPW
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: HemoSonics LLC (Industry)
Responsible Party: Principal Investigator, Bhavani Kodali, Director, University of Maryland, Baltimore
Other Study IDs: 84317
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hemorrhage; Coagulation Delay
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Pregnant Women: All subjects will have the same intervention. Samples will be taken and manipulated in the laboratory for use of the Hemosonic Qauntra Analyzer
  Interventions: Device: Quantra Analyzer

INTERVENTIONS:
Device: Quantra Analyzer — Subject's blood samples will be manipulated in the lab and will be tested with the Quantra Analyzer. After obtaining blood from each patient, the blood was diluted to varying dilutions to obtain different fibrinogen concentrations. This way, 89 samples were prepared from the blood from 13 patients. Each sample was analyzed for fibrinogen concentration in the lab using conventional technology. Additionally each sample was used to measure Quantra variables such as clot stiffness (CS), and fibrinogen contribution to clot stiffness (FCS).

SUMMARY:
In this study the investigators will evaluate a new point of care Quantra Hemostasis Analyzer system to assess coagulation rapidly with ease.

DETAILED DESCRIPTION:
Unexpected bleeding continues to be an issue that confronts anesthesiologists. Obstetric bleeding spearheads as the leading cause of maternal mortality and morbidity. One of the hurdles that clinicians confront is a lack of point of care coagulation system that can hasten the clinical management strategy in the right direction. Conventional methods take considerable time to obtain results. TEG and ROTEM are currently doing the job however these two modalities requires expertise and proficient training to perform test and interpret results. The level of expertise to run the TEG and ROTEM poses hurdles for providing coagulation around the clock as it requires trained operators. What is currently required for efficient and effective management of obstetric hemorrhage is a point of care coagulation system in the operating room and or labor and delivery suite that is user friendly, easy and quick to perform. In this study the investigators will evaluate a new point of care Quantra Hemostasis Analyzer system to assess coagulation rapidly with ease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman at 37-41 weeks gestation

Exclusion Criteria:

* Hypertension
* Preeclampsia
* Gestational diabetes
* Preexisting coagulopathy
* History of deep vein thrombosis (DVT)
* Medications that impair coagulation
* History of pulmonary embolism or thrombosis
* Women in active labor receiving intravenous fluids or oxytocin

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kodali, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kodali BS, Karuppiah A, Bharadwaj S, Chow J, Tanaka K. Efficacy of sonorheometry point of the care device in determining low fibrinogen levels in pregnant blood: an invitro dilution and reconstitution study. J Clin Monit Comput. 2022 Oct;36(5):1423-1431. doi: 10.1007/s10877-021-00782-1. Epub 2021 Dec 3. PMID 34859304

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women: All subjects will have the same intervention. Samples will be taken and manipulated in the laboratory for use of the Hemosonic Qauntra Analyzer
  Quantra Analyzer: Subjects blood will be manipulated in the lab and will be tested with the Quantra Analyzer
Period: Overall Study
Arm/Group | Pregnant Women
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant Women
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Hispanic or Non-Hispanic
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 13
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Fibrinogen in mg/dL Concentration With Clot Strength (CS hPa) and Fibrinogen Contribution to Clot (FCS hPa) of Point of the Care Quantra System.
Description: The Fibrinogen level of the patient in mg/dL is reflected by CS (clost strength measured in hPa) and FCS (Fibrinogen Contribution for Clot Stiffness measured by Quantra measured in hPa). CS and FCS are Quantra measurements of blood clot strength. The higher the CS and FCS, the stronger the clot and the higher the fibrinogen in the blood.
  Whole blood samples from pregnant women were diluted with saline to obtain various levels of fibrinogen. The diluted samples were reconstituted with plasma to obtain varying concentrations of fibrinogen. Each sample of the diluted and reconstituted blood was analyzed in the laboratory for fibrinogen level, as well as CS and FCS, using the Qunatra Point of Care system. The correlation between fibrinogen levels and respective CS and FCS was studied. The accuracy of FCS in determining low fibrinogen was the goal of the study. In all 89 samples were obtained from blood obtained from 13 participants.
Time Frame: Baseline: This is invitro study of the blood obtained from pregnant women (base line). This is a non-interventional observational study. Baseline samples were diluted and reconstituted and were analyzed on the same day within 4 hours of preparation.
Population: 89 samples were obtained from 13 subjects as explained above.
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: Samples
Groups:
- Fibrinogen Concentration in Each Sample: Blood obtained from pregnant patients served as baseline. The samples were diluted with saline and reconstituted with plasma to obtain varying levesl of fibrinogen. Fibrinogen was measured in the lab and Quantra Analyzer measured CS and FCS
Arm/Group | Fibrinogen Concentration in Each Sample
Number analyzed (Participants) | 13
Number analyzed (Samples) | 89
mg/dL
  Baseline values | 494 (103)
  Diluted with saline | 105 (31)
  15% reconstituted with non pregnant plasma | 137 (23)
  15% reconstituted with pregnant plasma | 162 (38)
  30% reconstituted with non pregnant plasma | 162 (25)
  30% reconstituted with pregnant plasma | 214 (46)
  Fully Resuscitated | 279 (38)
Statistical Analysis 1: Comparison: Fibrinogen Concentration in Each Sample; Using standard techniques for estimating sample size, a Delong's test indicated that a total of 61 samples would be sufcient to detect a 0.2 increase in the AUROC from the null hypothesis 0.5, assuming an alpha level of 5% and 90% power [12]. The manuscript was referenced against the STROBE checklist for cohort studies. Descriptive statistics were used to present; Test type: Other; p < 0.05, Regression, Linear; Correlation - R value = 0.93
Statistical Analysis 2: Comparison: Fibrinogen Concentration in Each Sample; Test type: Other; p < 0.05, Regression, Linear; Correlation - R value = 0.77

2. Primary Outcome: Correlation of Fibrinogen in mg/dL Concentration With Clot Strength (CS hPa) and Fibrinogen Contribution to Clot (FCS hPa) of Point of the Care Quantra System.
Description: The Fibrinogen level of the patient in mg/dL is reflected by CS (clot strength measured in hPa) and FCS (Fibrinogen Contribution for Clot Stiffness measured by Quantra measured in hPa). CS and FCS are Quantra measurements of blood clot strength. The higher the CS and FCS, the stronger the clot and the higher the fibrinogen in the blood.
  Whole blood samples from pregnant women were diluted with saline to obtain various levels of fibrinogen. The diluted samples were reconstituted with plasma to obtain varying concentrations of fibrinogen. Each sample of the diluted and reconstituted blood was analyzed in the laboratory for fibrinogen level, as well as CS and FCS, using the Qunatra Point of Care system. The correlation between fibrinogen levels and respective CS and FCS was studied. The accuracy of FCS in determining low fibrinogen was the goal of the study. In all 89 samples were obtained from blood obtained from 13 participants.
Time Frame: Baseline: This is invitro study of the blood obtained from pregnant women (base line). This is a non-interventional observational study. Baseline samples were diluted and reconstituted and were analyzed on the same day
Measure: Mean (Standard Deviation); unit: hPa
Units Other Than Participants: Samples
Groups:
- Quantra Measured Clot Stiffness CS; Quantra Measured FCS (Fibrinogen Contribution to Clot Strength: Blood obtained from pregnant patients served as baseline. The samples were diluted with saline and reconstituted with plasma.
Arm/Group | Quantra Measured Clot Stiffness CS | Quantra Measured FCS (Fibrinogen Contribution to Clot Strength
Number analyzed (Participants) | 13 | 13
Number analyzed (Samples) | 89 | 89
hPa
  Base line values | 32.8 (9.8) | 4.9 (2.5)
  Diluted with saline | 6.4 (2.2) | 1.1 (0.4)
  15% reconstituted with non pregnant plasma | 8.5 (1.6) | 1.9 (0.5)
  15% reconstituted with pregnant plasma | 10.9 (3.2) | 2.5 (0.9)
  30% reconstituted with non pregnant plasma | 8.8 (2.1) | 2.4 (0.8)
  30% reconstituted with pregnant plasma | 14.9 (4.5) | 3.8 (1.6)
  Fully resuscitated | 18.9 (4.5) | 3.9 (1.5)

ADVERSE EVENTS:
Time Frame: 2 days
Description: 0
Groups:
- Pregnant Women: All subjects will have the same intervention. Samples will be taken and manipulated in the laboratory for use of the Hemosonic Qauntra Analyzer Subjects had zero risk because the blood draws are from routine clinical draws. No additional risk involved because of the study.
  Quantra Analyzer: Subjects blood will be manipulated in the lab and will be tested with the Quantra Analyzer
Arm/Group | Pregnant Women
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Statistical data fibrinogen vs CS and FCS (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04301193/Prot_SAP_003.pdf
  • Informed Consent Form (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT04301193/ICF_002.pdf